CLINICAL TRIAL: NCT06335420
Title: Polyp Prophylactic Properties of Polyacetylenes in Patients With Previous Polypectomy
Brief Title: Prophylactic Properties of Carrot Juice in Patients With High-Risk Colorectal Polyps
Acronym: Px7
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Karolinska Institutet (Other); Umeå University (Other); Uppsala University Hospital (Other); Svendborg Hospital (Other); Ersta Hospital, Sweden (Other); St Goran's Hospital (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 324-2023-GB
Record Dates: First submitted 2024-03-13; First posted 2024-03-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer Prevention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carrot juice (Active Comparator): The cultivation of "Yellowstone" carrots will be conducted by DanRoots A/S.DanRoots, Organic Vegetables, Bjerringbro, Denmark.Juice is produced and taste corrected by Orskov Food, Denmark in collaboration with Naturfrisk, Ørbæk.
  Analysis of carrot juice for falcarinol and falcarindiol content will be done at random from 10 samples leaving the factory and 10 samples collected after 30 days storage at participant's homes for each batch.
  Interventions: Dietary Supplement: Carrot juice from Yellowstone carrots cultivars
- Placebo juice (Placebo Comparator): Placebo juice is produced from natural flavours and taste corrected by Orskov Food, Denmark in collaboration with Naturfrisk, Ørbæk. The taste is corrected to prevent enabling differentiation between carrot juice and placebo.
  Interventions: Dietary Supplement: Placebo juice

INTERVENTIONS:
Dietary Supplement: Carrot juice from Yellowstone carrots cultivars — Consumption of 100 ml of carrot juice daily for 1 year
  Arms: Carrot juice
Dietary Supplement: Placebo juice — Consumption of 100 ml of placebo juice daily for 1 year
  Arms: Placebo juice

SUMMARY:
The goal of this prospective randomized double-blinded bi-national study is to test the prophylactic effect of polyacetylenes from carrots on the population of patients who had a resection of high-risk adenomas of the large bowel.

The main question it aims to answer is: Will carrot juice rich in polyacetylenes inhibit neoplastic transformation and growth in high-risk humans?

Participants will have to drink 100 ml of juice daily after the adenoma resection for 1 year and keep a simple diary/calendar.

Researchers will compare the group with ingestion of Falcarinol (FaOH) / Falcarindiol (FaDOH) rich carrot juice versus the group consuming placebo juice, to see if the polyacetylenes significantly reduces neoplastic transformation and growth in high-risk patients.

DETAILED DESCRIPTION:
The study is a prospective double-blinded randomized controlled trial carried out in four centers: one Danish (Department of Surgery, Odense University Hospital - OUH) and five Swedish (Ersta Hospital - EH, Stockholm; Karolinska University Hospital - KUH, Stockholm; Uppsala University Hospital - UUH, Uppsala; Sahlgrenska University Hospital - SUH, Goteborg, Capio St. Gorans Hospital - CSH, Stockholm).

The investigators will organize two parallel arms of 400 patients: an intervention arm (consumption of 100 ml active carrot juice daily) and a control arm (consumption of 100 ml placebo juice daily) in a 1:1 randomized allocation ratio for 1 year. The project is structured in 2 working packages (WP):

1. The clinical trial (including cultivation and quality control of carrots and juice production; quantification of FaOH and FaDOH in the carrot and the placebo juice and the randomized trial)
2. The assessment of patient compliance and ways to improve it (Umeå Institute of Design, Umeå University - UMU).

The investigators hypothesize that the difference between the active arm (carrot juice) and the control arm (placebo juice) measured by number and growth rate (size) of recurrent adenomas will mediate a 20% reduction or larger in both size and number.

Outcomes will be investigated through standard colonoscopy report, questionnaires, calendars and diaries.

The randomization is stratified by inclusion center, each having its own block of 50/50 distribution between active and placebo arm.

The patients will collect 8 L of juice, the diary, calendar and a questionnaire every 2 months. At this meeting the patients will also have a follow-up discussion with the project nurse.

All patients will undergo colonoscopy after one year from the resection and in addition, for the piecemeal resections there will also be a local follow up colonoscopy after 6 months. Information about recurrence, the number of polyps, polyp size and characterization will be registered in the database. Full compliance is defined as consumption of > 75% of the juice delivered. Consumption data for all patients will be kept for compliance analysis.

Data will be analyzed using exact methods for binomial data. The combined endpoint will be the total number of recurrent adenomas multiplied with mean size of recurrent adenomas in the relevant treatment group.

Participation is voluntary with no economic compensation, and the patients are informed orally and in writing according to the information accepted by the ethics committee.

ELIGIBILITY:
Inclusion Criteria:

1. Any type of resection for adenomas larger than 20 mm in size (endoscopically evaluated) or endoscopically resected T1 cancers.
2. Acceptance of the treatment and follow-up program.
3. Capability to understand and follow the instructions.

Exclusion Criteria:

1. Patients allocated to "high-risk" group because of many small polyps (>4).
2. Pregnancy.
3. Known relevant allergies.
4. Chronic consumption of COX (cyclooxygenase) inhibitors (Aspirin, Celecoxib, Ibuprofen, Diclofenac, Ketoprofen, Ketorolac, Indometacin, Naproxen, Piroxicam) or immunosuppressive agents (Methotrexate, Azathioprine or glucocorticoids).
5. Patients with different neoplastic disease under treatment (Chemo-/Radio-/Imunotherapy).
6. Severe comorbidity NYHA III-IV.
7. Lynch syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Number and size of recurrent polyps found at the one-year follow up colonoscopy | 1 year
  The combined endpoint (number x size of recurrent polyps) after 1 year of treatment.

SECONDARY OUTCOMES:
Polyp number and mean size per patient and the relation with the carrot consumption measurement | 1 year
  A covariate analysis of carrot consumption (concentration of polyacetylenes exposure) measured through diaries, calendar and questionnaires and the findings at the 1 year colonoscopy (number of polyps multiplied by mean diameter of adenomas per patient).
Compliance rate (Juice consumption level) and side effects | 1 year
  Assessment of compliance rate and side effects through diary, calendar marks and questionnaire
The number of polyps with low, medium, high degree of dysplasia and cancer | 1 year
  Assessment of polyps through endoscopy and pathology reports
Acceptability of treatment | 1 year
  Assessment of acceptance and ways to improve carrot products through diary and questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Baatrup, Professor, Principal Investigator — OUH og Svendborg Sygehus
Locations (1):
- Department of Surgery, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deding U, Baatrup G, Kaalby L, Kobaek-Larsen M. Carrot Intake and Risk of Developing Cancer: A Prospective Cohort Study. Nutrients. 2023 Jan 29;15(3):678. doi: 10.3390/nu15030678. PMID 36771385
- [Background] Schmiech L. Strukturafklârung und qualitative Studien zu Bitterstoffen und Polyacetylenen in Karitten. Verlag Dr. Hut, 2011, ISBN 978-3-8439-0069-0
- [Background] Deding U, Clausen BH, Al-Najami I, Baatrup G, Jensen BL, Kobaek-Larsen M. Effect of Oral Intake of Carrot Juice on Cyclooxygenases and Cytokines in Healthy Human Blood Stimulated by Lipopolysaccharide. Nutrients. 2023 Jan 26;15(3):632. doi: 10.3390/nu15030632. PMID 36771338
- [Background] Jakobsen U, Kobaek-Larsen M, Kjoller KD, Antonsen S, Baatrup G, Trelle MB. Quantification of the anti-neoplastic polyacetylene falcarinol from carrots in human serum by LC-MS/MS. J Chromatogr B Analyt Technol Biomed Life Sci. 2022 Nov 1;1210:123440. doi: 10.1016/j.jchromb.2022.123440. Epub 2022 Sep 6. PMID 36088746
- [Background] Deding U, Baatrup G, Christensen LP, Kobaek-Larsen M. Carrot Intake and Risk of Colorectal Cancer: A Prospective Cohort Study of 57,053 Danes. Nutrients. 2020 Jan 27;12(2):332. doi: 10.3390/nu12020332. PMID 32012660
- [Background] Kobaek-Larsen M, Baatrup G, KhataeiNotabi M, El-Houri RB, Pipo-Olle E, Christensen Arnspang E, Christensen LP. Dietary Polyacetylenic Oxylipins Falcarinol and Falcarindiol Prevent Inflammation and Colorectal Neoplastic Transformation: A Mechanistic and Dose-Response Study in A Rat Model. Nutrients. 2019 Sep 14;11(9):2223. doi: 10.3390/nu11092223. PMID 31540047
- [Background] Kobaek-Larsen M, Nielsen DS, Kot W, Krych L, Christensen LP, Baatrup G. Effect of the dietary polyacetylenes falcarinol and falcarindiol on the gut microbiota composition in a rat model of colorectal cancer. BMC Res Notes. 2018 Jun 27;11(1):411. doi: 10.1186/s13104-018-3527-y. PMID 29945666
- [Background] Kobaek-Larsen M, El-Houri RB, Christensen LP, Al-Najami I, Frette X, Baatrup G. Dietary polyacetylenes, falcarinol and falcarindiol, isolated from carrots prevents the formation of neoplastic lesions in the colon of azoxymethane-induced rats. Food Funct. 2017 Mar 22;8(3):964-974. doi: 10.1039/c7fo00110j. PMID 28197615
- [Background] Kobaek-Larsen M, Christensen LP, Vach W, Ritskes-Hoitinga J, Brandt K. Inhibitory effects of feeding with carrots or (-)-falcarinol on development of azoxymethane-induced preneoplastic lesions in the rat colon. J Agric Food Chem. 2005 Mar 9;53(5):1823-7. doi: 10.1021/jf048519s. PMID 15740080
- [Derived] Agache A, Deding U, Kaalby L, Kobaek-Larsen M, Al-Najami I, Ostergaard Hansen L, Stryhn C, Wilde D, Forsberg A, Backman AS, Bates T, de Lange T, Martling A, Baatrup G. Polyp prophylactic properties of polyacetylenes from carrots in patients with previous polypectomy-Px7 The study protocol of a multicentre binational randomised controlled trial. BMJ Open. 2025 Nov 28;15(11):e095376. doi: 10.1136/bmjopen-2024-095376. PMID 41314836

DOCUMENTS (2):
  • Study Protocol (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT06335420/Prot_000.pdf
  • Informed Consent Form (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT06335420/ICF_001.pdf